CLINICAL TRIAL: NCT03715673
Title: Von Willebrand Antigen and Activity as Novel Biomarkers of Hemostasis in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Abozied Abdallah, clinical hematology specialist, Assiut University
Other Study IDs: vWF in IBD
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Inflammatory Bowel Diseases; Von Willebrand Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; von Willebrand Diseases | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases:Active IBD patients: 23 patients with active inflammatory bowel disease for whom von willlebrand antigen and activity will be done
  Interventions: Diagnostic Test: von willebrand antigen and activity
- Control:Inactive IBD patients: 23 patients with inactive inflammatory bowel disease; VWF antigen and activity will be done for them
  Interventions: Diagnostic Test: von willebrand antigen and activity

INTERVENTIONS:
Diagnostic Test: von willebrand antigen and activity — Measuring von Willebrand antigen and activity (VWF: RCo and VWF: CB)

SUMMARY:
The investigators are going to study von Willebrand antigen and activity levels in patients with inflammatory bowel disease. The study will be on 46 patients who were diagnosed with inflammatory bowel disease mainly ulcerative colitis and Crohn's disease divided into two arms; group A will include 23 cases with active IBD(cases)status and group B will include 23 cases with inactive IBD status(control) to compare the vWF antigen and activity ( expected to be higher in active disease group.

The investigators will follow all of the patients for any arterial or venous thrombosis to evaluate IBD as a risk factor of thrombosis, on the other hand, they are looking to detect cases of acquired von Willebrand syndrome in some cases with bleeding that not explained by the inflammatory bowel disease status.

The aim of the work:

1. Assessment of VWF antigen in patients with inflammatory bowel disease and correlate it to disease activity.
2. Evaluation of VWF antigen as a risk factor for thrombosis in inflammatory bowel disease patients.
3. Detection of acquired von Willebrand disease in inflammatory bowel disease.

DETAILED DESCRIPTION:
VWF is a high-molecular-weight multimeric glycoprotein, synthesized and released by vascular endothelial cells and megakaryocytes that play an important role in platelet-endothelial cell interaction and stabilizing the factor VIII (FVIII) coagulation protein.

Von Willebrand factor (VWF) is an acute-phase protein and a marker of endothelial damage.

VWF is crucial for platelet adhesion and aggregation. High-molecular weight multimers (HMWMs) are involved in platelet aggregation under high shear stress but under normal conditions it presents solely in the subendothelium and released into the bloodstream following activation of endothelial cells.

Coagulation and inflammation are simultaneously activated and respond in synergy as a preserved mechanism to repair the injured areas during tissue damage.

This observation is particularly relevant in acute inflammatory diseases, such as sepsis, but it also seems to be very important in chronic inflammatory conditions, such as inflammatory bowel disease.

Inflammatory bowel disease (IBD) with its two main forms, ulcerative colitis (UC) and Crohn disease (CD), is a chronic inflammatory condition characterized by local and systemic inflammation predominantly affecting the gastrointestinal tract and well known to be associated with a hypercoagulable state and subsequently with an increased risk for venous thromboembolism (VTE).

Thromboembolic complications such as Deep Venous Thrombosis (DVT) and Pulmonary Embolism (PE) represent amongst IBD complications an important and underestimated factor to be borne in mind which can significantly influence patient's morbidity and mortality.

In fact, according to the latest population-cohort studies, a 2 to 3-time fold increased risk of developing of thromboembolic complications was reported for IBD patients compared to general population.

In particular as Grainge., et al. and Papa., et al. both demonstrate in their studies, the incidence of thromboembolic events varies depending on the activity phase of the disease, suggesting that there is a higher risk of thromboembolic complications especially during IBD flares, with similar relative risk values for both Crohn's Disease and Ulcerative Colitis.

Although the causes of the increased risk of VTE in IBD are not yet completely understood, endothelial dysfunction has been demonstrated in IBD and it is evident through increasing levels of endothelial injury markers. The most frequently used biochemical markers of endothelial damage include von Willebrand factor (vWF), TM, vascular cell adhesion molecule 1 (VCAM-1), intercellular adhesion molecule 1 (ICAM-1) and endothelin-1 (ET-1).

In 2017 Cibor et al published the first report of the effects of parameters associated with the structure and function of VWF on hemostasis in IBD. On the one hand, ADAMTS13: Ag was lower in IBD patients than in controls, particularly in subjects with UC; this resulted in an increased number of circulating multimers of VWF and thus an elevated thrombotic risk. The prothrombotic effects are enhanced by markedly elevated VWF: Ag.

On the other hand, the incidence of AVWS, which leads to an increased risk for bleeding, was higher in IBD patients. These findings provide insight into the elevated risk for thromboembolic events and bleeding observed in UC and less frequently in CD. The dysregulation of the balance between VWF function and ADAMTS13 reported herein might contribute to the complex hemostatic abnormalities observed in IBD.

Currently, the association between CD and AVWS is likely underestimated, especially in cases of acute bleeding not related to disease activity.

In 2017 Di Sabatino, et al reported three cases of IBD patients, who developed severe hemorrhagic manifestations due to the concomitant presence of an AVWS, in addition to other three cases was described in the literature. Such a condition can be life-threatening and its timely identiﬁcation is mandatory to adopt the optimal therapeutic strategy.

The association between AVWS and IBD might be more frequent than expected. The autoimmune pathogenesis of IBD makes the association more likely. The availability of specialized coagulation centers and correlation with clinical information should confirm the diagnosis.

Methodology:

Patients will be subjected to the following:

Clinical assessment:

1. The clinical assessment will include demographic data, the presence of comorbidities, cigarette-smoking habits, previous history of thromboembolism and medications.
2. Body mass index (BMI) will be calculated for all patients.
3. In patients with CD and UC, the following parameters will be evaluated: disease duration, disease location, disease activity, complications, and past surgical procedures. Complications are defined as abscesses, fistulae, and stenoses.
4. Disease activity will be assessed according to ECCO-ESGAR Consensus Guidelines 2018.

Laboratory assessment:

The following will be done for all patients:

1. WBC, hematocrit, platelet count.
2. partial activated thromboplastin time.
3. C-reactive protein (CRP), and fecal calprotectin.
4. VWF: Ag, VWF: RCo and VWF: CB.

Radiological tests:

In cases with suspected arterial or venous thromboembolism, the appropriate radiological study will be done (i.e. venous doppler for deep venous thrombosis).

ELIGIBILITY:
Inclusion Criteria:

•Patients with inflammatory bowel disease either newly or previously diagnosed aged18 years and older.

Exclusion Criteria:

* Pregnancy.
* Myocardial infarction.
* Stroke.
* Thromboembolism.
* Known hemorrhagic diathesis.
* Cancer.
* Renal insufficiency.
* Liver injury.
* Diabetes.
* patients who are on aspirin, heparin, oral anticoagulants, or oral contraceptives pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with inflammatory bowel disease either newly or previously diagnosed aged 18 years and older following in Assiut university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
comparison of von willebrand antigen and activity between the two groups | baseline
  Assessment of von willebrand antigen level as an activity marker in inflammatory bowel disease patients.
detection of arterial or venous thrombosis | follow up for one year
  all patients will be followed for detection of any thrombotic events to evaluate the thrombotic risk in IBD
detection of acquired von willebrand syndrome | follow up for one year
  All patients who have bleeding not explained by the IBD status will be investigated for detection of any cases of acquired von willebrand syndrome.

SECONDARY OUTCOMES:
Estimation of the prevalence of IBD patients attending our clinic (Assiut University Experience). | one year
  prevalence of inflammatory bowel disease in assiut university hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Yee A, Kretz CA. Von Willebrand factor: form for function. Semin Thromb Hemost. 2014 Feb;40(1):17-27. doi: 10.1055/s-0033-1363155. Epub 2013 Dec 13. PMID 24338608
- [Background] Cibor D, Domagala-Rodacka R, Rodacki T, Jurczyszyn A, Mach T, Owczarek D. Endothelial dysfunction in inflammatory bowel diseases: Pathogenesis, assessment and implications. World J Gastroenterol. 2016 Jan 21;22(3):1067-77. doi: 10.3748/wjg.v22.i3.1067. PMID 26811647
- [Background] Reininger AJ. The function of ultra-large von Willebrand factor multimers in high shear flow controlled by ADAMTS13. Hamostaseologie. 2015;35(3):225-33. doi: 10.5482/HAMO-14-12-0077. Epub 2015 May 18. PMID 25983111
- [Background] Lipinski S, Bremer L, Lammers T, Thieme F, Schreiber S, Rosenstiel P. Coagulation and inflammation. Molecular insights and diagnostic implications. Hamostaseologie. 2011 May 2;31(2):94-102, 104. doi: 10.5482/ha-1134. Epub 2010 Dec 9. PMID 21152678
- [Background] Esmon CT. The interactions between inflammation and coagulation. Br J Haematol. 2005 Nov;131(4):417-30. doi: 10.1111/j.1365-2141.2005.05753.x. PMID 16281932
- [Background] Owczarek D, Cibor D, Glowacki MK, Rodacki T, Mach T. Inflammatory bowel disease: epidemiology, pathology and risk factors for hypercoagulability. World J Gastroenterol. 2014 Jan 7;20(1):53-63. doi: 10.3748/wjg.v20.i1.53. PMID 24415858
- [Background] Arora Z, Wu X, Navaneethan U, Shen B. Non-surgical porto-mesenteric vein thrombosis is associated with worse long-term outcomes in inflammatory bowel diseases. Gastroenterol Rep (Oxf). 2016 Aug;4(3):210-5. doi: 10.1093/gastro/gov012. Epub 2015 Apr 28. PMID 25922204
- [Background] Bollen L, Vande Casteele N, Peeters M, Van Assche G, Ferrante M, Van Moerkercke W, Declerck P, Vermeire S, Gils A. The Occurrence of Thrombosis in Inflammatory Bowel Disease Is Reflected in the Clot Lysis Profile. Inflamm Bowel Dis. 2015 Nov;21(11):2540-8. doi: 10.1097/MIB.0000000000000531. PMID 26313696
- [Background] Grainge MJ, West J, Card TR. Venous thromboembolism during active disease and remission in inflammatory bowel disease: a cohort study. Lancet. 2010 Feb 20;375(9715):657-63. doi: 10.1016/S0140-6736(09)61963-2. Epub 2010 Feb 8. PMID 20149425
- [Background] Papa A, Gerardi V, Marzo M, Felice C, Rapaccini GL, Gasbarrini A. Venous thromboembolism in patients with inflammatory bowel disease: focus on prevention and treatment. World J Gastroenterol. 2014 Mar 28;20(12):3173-9. doi: 10.3748/wjg.v20.i12.3173. PMID 24695669
- [Background] Cromer WE, Mathis JM, Granger DN, Chaitanya GV, Alexander JS. Role of the endothelium in inflammatory bowel diseases. World J Gastroenterol. 2011 Feb 7;17(5):578-93. doi: 10.3748/wjg.v17.i5.578. PMID 21350707
- [Background] Cibor D, Owczarek D, Butenas S, Salapa K, Mach T, Undas A. Levels and activities of von Willebrand factor and metalloproteinase with thrombospondin type-1 motif, number 13 in inflammatory bowel diseases. World J Gastroenterol. 2017 Jul 14;23(26):4796-4805. doi: 10.3748/wjg.v23.i26.4796. PMID 28765701
- [Background] Di Sabatino A, Ambaglio C, Aronico N, Ghidelli N, Lenti MV, Gamba G, Corazza GR. Acquired von Willebrand syndrome in inflammatory bowel disease. Haemophilia. 2017 May;23(3):e231-e233. doi: 10.1111/hae.13209. Epub 2017 Mar 17. No abstract available. PMID 28314057
- [Background] Federici AB, Budde U, Castaman G, Rand JH, Tiede A. Current diagnostic and therapeutic approaches to patients with acquired von Willebrand syndrome: a 2013 update. Semin Thromb Hemost. 2013 Mar;39(2):191-201. doi: 10.1055/s-0033-1334867. Epub 2013 Feb 8. PMID 23397553